CLINICAL TRIAL: NCT02585713
Title: A Phase III, Randomized, Open Label Study Evaluating the Safety of Apixaban in Subjects With Cancer Related Venous Thromboembolism
Brief Title: Apixaban or Dalteparin in Reducing Blood Clots in Patients With Cancer Related Venous Thromboembolism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RU221501I; NCI-2015-01573 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CV185-444; RU221501I (Other: Academic and Community Cancer Research United)
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2019-06

CONDITIONS: Cerebral Vein Thrombosis; Deep Vein Thrombosis; Gonadal Thrombosis; Hepatic Thrombosis; Malignant Neoplasm; Mesenteric Thrombosis; Metastatic Malignant Neoplasm; Portal Vein Thrombosis; Pulmonary Embolism; Renal Vein Thrombosis; Splenic Thrombosis; Venous Thromboembolism
MeSH Terms: conditions — Intracranial Thrombosis; Venous Thrombosis; Neoplasms; Mesenteric Ischemia; Neoplasm Metastasis; Pulmonary Embolism; Venous Thromboembolism | interventions — apixaban; Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (apixaban) (Experimental): Patients receive apixaban 10 mg PO BID on days 1-7 and lower-dose apixaban 5 mg PO BID on days 8-180.
  Interventions: Drug: Apixaban; Other: Questionnaire Administration
- Arm II (dalteparin) (Experimental): Patients receive dalteparin 200 IU/kg/day SC QD on days 1-30 and lower-dose dalteparin 150 IU/kg/day SC QD on days 31-180.
  Interventions: Drug: Dalteparin; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Apixaban — Given PO
  Other Names: BMS-562247; BMS-562247-01; Eliquis
  Arms: Arm I (apixaban)
Drug: Dalteparin — Given SC
  Arms: Arm II (dalteparin)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies the side effects of and compares apixaban and dalteparin in reducing blood clots in patients with cancer-related venous thromboembolism. Venous thromboembolism is a condition in which a blood clot forms in a vein and then breaks off and moves through the bloodstream. Patients with cancer are at increased risk for venous thromboembolism. Apixaban and dalteparin are drugs used to prevent blood clots from forming or to treat blood clots that have formed. It is not yet known whether apixaban or dalteparin is more effective in reducing blood clots in patients with cancer related venous thromboembolism.

ADAM-VTE

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Any episode of major bleeding including fatal bleeding.

SECONDARY OBJECTIVES:

I. Venous thromboembolism (VTE) recurrence including deep vein thrombosis (DVT), pulmonary embolism (PE), fatal PE, or arterial thromboembolism.

II. Any episode of major bleeding including fatal bleeding or any episode of clinically relevant non-major bleeding.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive apixaban 10 mg orally (PO) twice daily (BID) on days 1-7 and lower-dose apixaban 5 mg PO BID on days 8-180.

ARM II: Patients receive dalteparin 200 international units (IU)/kg/day subcutaneously (SC) once daily (QD) on days 1-30 and lower-dose dalteparin 150 IU/kg/day SC QD on days 31-180.

After completion of study treatment, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute lower extremity or upper extremity (jugular, innominate, subclavian, axillary, brachial) DVT, PE, splanchnic (hepatic, portal, splenic, mesenteric, renal, gonadal), or cerebral vein thrombosis
* Active cancer defined as metastatic disease and/or any evidence of cancer on cross-sectional or positron emission tomography (PET) imaging, cancer related surgery, chemotherapy or radiation therapy within the past 6 months; note: non-melanoma skin cancer does not meet the cancer requirement
* Life expectancy >= 60 days
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Obtained =< 30 days prior to randomization: Platelet count >= 50,000/mm^3
* Obtained =< 30 days prior to randomization: Alanine aminotransferase (ALT) or aspartate transaminase (AST) =< 3 x upper limit of normal (ULN)
* Obtained =< 30 days prior to randomization: International normalized ratio (INR) =< 1.6 (if not taking anticoagulant therapy)
* Obtained =< 30 days prior to randomization: Calculated creatinine clearance must be >= 30 ml/min using the Cockcroft-Gault formula
* Negative serum or urine pregnancy test done =< 24 hours prior to randomization, for women of childbearing potential only; note: a women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal; menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes
* Ability to complete questionnaire(s) by themselves or with assistance
* Ability to provide informed written consent
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

    * Note: women of child bearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 33 days after finishing the last dose
    * Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 93 days after finishing the last dose
    * Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements; however they must still undergo pregnancy testing as described in this section
* Note: investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception; highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly
* At a minimum, subjects must agree to the use of one method of highly effective contraception as listed below:

  * HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

    * Male condoms with spermicide
    * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject?s WOCBP partner
    * Female partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
    * IUDs, such as ParaGard
    * Tubal ligation
    * Vasectomy
    * Complete abstinence

      * Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs; female subjects must continue to have pregnancy tests; acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence
* Treatment with an anticoagulant for more than 7 days for the current blood clot, prior to randomization
* Active bleeding
* Severe hypersensitivity reaction to apixaban, dalteparin, heparin or pork products (e.g., anaphylactic reactions)
* Use of the following CYP3A4 inducers: rifampin, rifabutin, carbamazepine, efavirenz, phenobarbital, phenytoin, fosphenytoin, primidone, and St. John?s wort)
* Thienopyridine therapy (clopidogrel, prasugrel, or ticagrelor) that will be continued on study
* Severe liver disease (known cirrhosis Childs Pugh class B or C), or active hepatitis
* Use of a Factor Xa inhibitor (e.g. apixaban, rivaroxaban, or edoxaban) =< 3 months prior to randomization
* Treatment of a thromboembolic event =< 6 months prior to randomization
* Documented venous thromboembolism while on therapeutic anticoagulation (?anticoagulation failure?)
* Mechanical heart valve
* Documented hemorrhagic tendencies
* Bacterial endocarditis
* History of heparin induced thrombocytopenia
* Any of the following conditions:

  * Intracranial bleeding =< 6 months prior to randomization
  * Intraocular bleeding =< 6 months prior to randomization
  * Gastrointestinal bleeding and/or endoscopically proven ulcer =< 6 months prior to randomization
  * Head trauma or major trauma =<1 month prior to randomization
  * Neurosurgery =< 2 weeks prior to randomization
  * Major surgery =< 1 week prior to randomization
  * Overt major bleeding at the time of randomization
  * Gross hematuria at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2019-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McBane, Principal Investigator — Academic and Community Cancer Research United
Locations (18):
- United States (18):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota

REFERENCES:
- [Derived] McBane RD 2nd, Wysokinski WE, Le-Rademacher JG, Zemla T, Ashrani A, Tafur A, Perepu U, Anderson D, Gundabolu K, Kuzma C, Perez Botero J, Leon Ferre RA, Henkin S, Lenz CJ, Houghton DE, Vishnu P, Loprinzi CL. Apixaban and dalteparin in active malignancy-associated venous thromboembolism: The ADAM VTE trial. J Thromb Haemost. 2020 Feb;18(2):411-421. doi: 10.1111/jth.14662. Epub 2019 Nov 28. PMID 31630479
- [Derived] McBane Ii R, Loprinzi CL, Ashrani A, Perez-Botero J, Leon Ferre RA, Henkin S, Lenz CJ, Le-Rademacher JG, Wysokinski WE. Apixaban and dalteparin in active malignancy associated venous thromboembolism. The ADAM VTE Trial. Thromb Haemost. 2017 Oct 5;117(10):1952-1961. doi: 10.1160/TH17-03-0193. Epub 2017 Aug 24. PMID 28837207

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Apixaban): Patients receive apixaban 10 mg PO BID on days 1-7 and lower-dose apixaban 5 mg PO BID on days 8-180.
- Arm B (Dalteparin): Patients receive dalteparin 200 IU/kg/day SC QD on days 1-30 and lower-dose dalteparin 150 IU/kg/day SC QD on days 31-180.
Period: Overall Study
Arm/Group | Arm A (Apixaban) | Arm B (Dalteparin)
Started | 150 | 150
Completed (Received Treatment; Primary Analysis Population) | 145 | 142
Not Completed | 5 | 8
Not completed — Withdrew prior to treatment | 2 | 7
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Apixaban) | Arm B (Dalteparin) | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (11.3) | 64.0 (10.8) | 64.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 77 | 155
  Male | 72 | 73 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 11 | 17
  White | 140 | 138 | 278
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 60 | 62 | 122
    1 | 70 | 76 | 146
    2 | 20 | 12 | 32

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Bleeding Rate
Description: The rate (percentage) of patients experiencing major bleeding at 6 months from treatment initiation and its associated 95% confidence interval was estimated separately by treatment arm using a cumulative incidence function, treating death without bleeding as a competing risk.
Time Frame: Up to 6 months
Population: Primary Analysis Population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Apixaban) | Arm B (Dalteparin)
Number analyzed (Participants) | 145 | 142
percentage of patients | 0 [0 to 0] | 2.1 [0.6 to 6.6]

2. Secondary Outcome: Composite Bleeding Rate: Major Bleed or a Clinically Relevant Non-major Bleed
Description: A similar analysis as described for the primary safety analysis will be used. The rate (percentage) of patients experiencing major bleeding or a clinically relevant non-major bleed at 6 months from treatment initiation and its associated 95% confidence interval was estimated separately by treatment arm using a cumulative incidence function, treating death without bleeding as a competing risk.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Apixaban) | Arm B (Dalteparin)
Number analyzed (Participants) | 145 | 142
percentage of patients | 7.0 [4.1 to 11.9] | 8.1 [4.7 to 13.9]

3. Secondary Outcome: Time to the First Event of the Composite Deep Vein Thrombosis (DVT)/Pulmonary Embolism (PE)
Description: Analyzed using the same methods described above for the primary endpoint.Time to the first event of the composite deep vein thrombosis (DVT)/pulmonary embolism (PE) is defined as the time from randomization to the date the patient experienced the first event of the composite deep vein thrombosis (DVT)/pulmonary embolism (PE).
Time Frame: Up to 3 months post-treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Apixaban) | Arm B (Dalteparin)
Number analyzed (Participants) | 149 | 149
months | NA [NA to NA] — The median and 95% CI was not reached due to limited number of events. | NA [NA to NA] — The median and 95% CI was not reached due to limited number of events.
Statistical Analysis 1: Comparison: Arm A (Apixaban) vs Arm B (Dalteparin); Test type: Superiority; p = 0.1316, Log Rank

ADVERSE EVENTS:
Time Frame: Up to 3 months after completion of treatment
Description: Adverse events are summarized below for patients who received at least one cycle of treatment (i.e. patients who completed the study and patients with unknown reason for not completing the study in the Participant Flow) and completed at least one adverse event form.
Arm/Group | Arm A (Apixaban) | Arm B (Dalteparin)
All-Cause Mortality (participants affected / at risk) | 35/148 | 25/143
Serious Adverse Events (participants affected / at risk) | 62/148 | 51/143
Other Adverse Events (participants affected / at risk) | 78/148 | 71/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Apixaban) (N=148) | Arm B (Dalteparin) (N=143)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (2)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Duodenal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 3 (3)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 3 (3)
Death NOS (General disorders) | 3 (3) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 2 (3)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (2)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Esophageal infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 3 (4)
Lung infection (Infections and infestations) | 5 (5) | 3 (4)
Sepsis (Infections and infestations) | 1 (1) | 5 (6)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (2)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 3 (3)
INR increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (3) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 32 (35) | 24 (26)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 2 (2)
Fallopian tube obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 2 (2) | 7 (7)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Apixaban) (N=148) | Arm B (Dalteparin) (N=143)
Anemia (Blood and lymphatic system disorders) | 14 (28) | 12 (22)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 3 (3)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 29 (70)
Pain (General disorders) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bone infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (2) | 0 (0)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 2 (2)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Alkaline phosphatase increased (Investigations) | 3 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 2 (3)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 2 (2)
INR increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 9 (18) | 8 (13)
Lymphocyte count increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 10 (16) | 7 (23)
Platelet count decreased (Investigations) | 40 (93) | 26 (71)
Weight gain (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 2 (3) | 1 (1)
White blood cell decreased (Investigations) | 7 (16) | 7 (21)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 4 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (5) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bleeding (Vascular disorders) | 31 (38) | 23 (27)
Hypertension (Vascular disorders) | 5 (9) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT02585713/Prot_SAP_000.pdf